CLINICAL TRIAL: NCT00081003
Title: The Intraduct Environment: A Novel Approach to Risk Assessment of Women With a Family History of Breast Cancer
Brief Title: Nipple Aspiration, Ductal Lavage, and Duct Endoscopy in Screening Women at Moderate-to-High Risk of Developing Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Screening
Other Study IDs: CDR0000358797; RMNHS-2278; EU-20352
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2005-12

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gene Expression Profiling; Endoscopic Mucosal Resection

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: protein expression analysis
Other: cytology specimen collection procedure
Other: laboratory biomarker analysis
Other: physiologic testing
Procedure: breast duct lavage
Procedure: endoscopic biopsy
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Screening tests, such as nipple aspiration, ductal lavage, and breast duct endoscopy, may help doctors detect cancer cells early and plan more effective treatment for breast cancer.

PURPOSE: This clinical trial is studying how well nipple aspiration, ductal lavage, and breast duct endoscopy work in detecting cancer cells in healthy women who are at moderate-to-high risk of developing breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the incidence of mild or severe cellular atypia in nipple aspirate fluid of healthy women at moderate to high risk of developing breast cancer, defined by family history or prior atypical biopsy.

Secondary

* Correlate cellular atypia with breast cancer, biochemical tumor markers, growth factors, and genetic and protein markers in these participants.
* Determine cancer risk and incidence utilizing these methods of screening in these participants.
* Observe the natural history of atypia in these participants over a total of 10 years.
* Determine whether these techniques may serve as supplementary tools in future screening of these participants.

OUTLINE: Participants under 50 years of age undergo nipple aspiration every twelve months for 3 years. Participants over 50 years of age undergo nipple aspiration every 18 months for 4.5 years.

Participants with significant cellular atypia in nipple aspirate fluid undergo ductal lavage and endoscopy.

Participants are followed annually for a total of 10 years.

PROJECTED ACCRUAL: A total of 1,000 participants will be accrued for this study within approximately 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Significant family history or prior atypical biopsy indicative of a moderate or high risk of developing breast cancer
* No concurrent inflammatory breast cancer
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 to 64

Sex

* Female

Menopausal Status

* Premenopausal or postmenopausal

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No prior allergy to EMLA cream or lidocaine
* No severe illness that would preclude study participation
* No mental illness or handicap that would preclude study compliance
* No concurrent active infection or inflammation in the breast being studied
* Not unconscious
* Not pregnant
* No nursing within the past 12 months

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* No prior subareolar surgery (e.g., microdochectomy or major duct excision) that may disrupt the ductal systems within 2 cm of the nipple
* No prior breast implantation on proposed lavage side

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2003-11

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Gui, MD, MS, FRCS(Edin), FRCS(Eng), Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden - London, London, England, United Kingdom